CLINICAL TRIAL: NCT01497678
Title: Musculotendinous Tissue Unit Repair and Reinforcement (MTURR) With the Use of Biologic Scaffolds for Patients Suffering From Severe Skeletal Muscle Injury (Coordinating Center Protocol)
Brief Title: Musculotendinous Tissue Unit Repair and Reinforcement (MTURR) Coordinating Center
Acronym: MTURR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues. 0 subjects enrolled
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11050209
Record Dates: First submitted 2011-08-09; First posted 2011-12-22 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Traumatic Injury; Muscle Injury; Tendon Injury; Soft Tissue Injury; Extremity Injury
Keywords: MTURR; ECM; Muscle Loss; Tendon; Tendon Repair; Muscle Repair; Soft Tissue Repair; Scaffold; Extracellular Matrix
MeSH Terms: conditions — Wounds and Injuries; Tendon Injuries; Soft Tissue Injuries; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extracellular Matrix (Other): Implantation of Extracellular Matrix
  Interventions: Device: Extracellular Matrix

INTERVENTIONS:
Device: Extracellular Matrix — Extracellular Matrix

SUMMARY:
The objective of the study is to assess mechanical strength and function in subjects undergoing Musculotendinous Tissue Unit Repair and Reinforcement (MTURR) with the use of biologic scaffolds for the restoration of both mechanical strength and function in these subjects. This study will formally evaluate healing and return of function after an extracellular matrix device implantation in 40 male and female subjects participating at 4-5 military sites who suffer from injury with loss of skeletal muscle tissue. The University of Pittsburgh under the Department of Plastic and Reconstructive Surgery is the Coordinating Center for this multi-site study.

DETAILED DESCRIPTION:
Loss of musculotendinous tissue as a result of trauma inevitably leads to severe morbidity for the subject and surgical challenges for the caregiver. The reconstruction of tissue following such injuries is often not possible and surgical options are extremely limited. Amputation of the affected limb is not an uncommon outcome. Free muscle grafts, pedicle grafts, and the use of prosthetic materials have all been attempted when primary repair is not possible due to loss of tissue domain. The results of such efforts are typically disheartening. If autologous grafts are used, donor site morbidity compounds the post surgical problems with resultant diminished quality of life. Stated differently, the existing treatment options for treatment of the loss of large amounts of skeletal muscle tissue with scarring are extremely limited because the existing tendon structures are damaged and lack strength. A Repair and Reinforcement approach with a biocompatible device would represent a paradigm shift in the treatment of traumatic tissue injury. This approach involves releasing scar tissue that constricts movement of the existing tendon, repairing damaged tendon and musculotendinous units with suture repair, and reinforcing the repair with a biologic scaffold material. The biologic scaffold is composed of animal derived collagen and the approved by the FDA as devices for reinforcement of soft tissues repaired by sutures or suture anchors, during tendon repair surgery." Additionally, as listed in the FDA 510k approval, these devices" provide a remodelable scaffold that is replaced by the subject's own soft tissues." These biologic materials fall into a category of implantable devices known as extracellular matrix (ECM) because they are composed of proteins that surround the cellular elements in mammals. No living cells are found in these ECM implantable devices. ECM devices are made by many commercial manufacturers and have been used for a variety of reconstructive surgical procedures for years. Because the ECM implant becomes populated with subject cells and blood vessels, the repair may be stronger and the new tissue growing within the device could possibly contribute to improved function by augmenting the tendon structure and allowing ingrowth of adjacent muscle fibers. The objective of the study is to assess mechanical strength and function in subjects undergoing Musculotendinous Tissue Unit Repair and Reinforcement (MTURR) with the use of biologic scaffolds for the restoration of both mechanical strength and function in these subjects. This study will formally evaluate healing and return of function after an extracellular matrix device implantation in 40 male and female subjects participating at 4-5 military sties who suffer from injury with loss of skeletal muscle tissue. The University of Pittsburgh under the Department of Plastic Surgery is the Coordinating Center for this multi-site study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following characteristics will be eligible to participate in the study:

  * Age: 18 to 70 years of age and able to provide informed consent
  * Civilian, and current or former military personnel are eligible to participate
  * Have suffered injury resulting in a structural deficit of a minimum of 20% of the muscle group mass and a functional deficit of a minimum of 25% when compared to the contralateral limb; or if bilateral injury is present to extremities, the potential surgical extremity is to be compared against normal expected values of a sample population of similar age and gender, and evidence of remaining tendon and musculotendinous units that could be surgically repaired with sutures.
  * Injuries may encompass a single muscle belly or compartment. Whether an area is expected to be repaired by sutures will be determined from imaging studies and physical examination.
  * Have suffered traumatic injury within the last 18 months to the upper and/or lower extremity; Target of 18 months or less but subject's may be enrolled with injury outside this range if the principal investigator determines that there is viable muscle in the injured compartment determined by clinical exam and imaging studies.
  * Eligible for study procedures 3 months post injury with stability determined by the Principal Investigator and/ or MD Co-Investigator
  * Willing and able to comply with follow up examinations, radiographic studies, physical therapy, muscle biopsy and laboratory tests.

Exclusion Criteria:

* Patients with the following characteristics will be excluded from participating in the study:

  * Inability to provide informed consent
  * Poor nutrition (demonstrated by abnormal lab range for serum Albumin and Pre-Albumin values)
  * Chronic disease such as congestive heart failure, liver disease, renal disease, or diabetes
  * Active and unstable disease state or infection anywhere in the body per MD's evaluation and determination (demonstrated by stated or medical record history and abnormal lab range for CBC with Differential and Platelet, and chemistry panel values)
  * Known coagulopathy (demonstrated by stated or medical record history of diagnosis)
  * Pregnancy (demonstrated by a positive result of a urine pregnancy test)
  * Diagnosis of cancer within last 12 months and /or actively receiving chemotherapy or radiation treatment
  * Axis I diagnosis DSM-IV (e.g., Schizophrenia, Bipolar Disorder). Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion
  * Subjects with complete muscle/tendon gaps greater than 5 cm that are obvious on imaging studies and are unlikely to be reasonably repaired with sutures and reinforcement, and will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mechanical strength and function | Approximately 6 months post-operative
  The primary objective of the study is to assess mechanical strength and function of surgical extremity in patients undergoing Musculotendinous Tissue Unit Repair and Reinforcement (MTURR) with the use of biologic scaffolds for the restoration of both mechanical strength and function in these patients. Physical therapy evaluations of strength and active/passive range of motion and self-reported measures of ability to perform activities of daily living.

SECONDARY OUTCOMES:
Pathology Evaluation | Approximately 6 months post-operative
  The secondary objective is to examine the cellular properties of the biopsy tissue material from the Extracellular Matrix surgical site for reabsorption and replacement by the subjects own soft tissue with pathological findings to be correlated with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Valentin JE, Badylak JS, McCabe GP, Badylak SF. Extracellular matrix bioscaffolds for orthopaedic applications. A comparative histologic study. J Bone Joint Surg Am. 2006 Dec;88(12):2673-86. doi: 10.2106/JBJS.E.01008. PMID 17142418
- [Background] Beattie AJ, Gilbert TW, Guyot JP, Yates AJ, Badylak SF. Chemoattraction of progenitor cells by remodeling extracellular matrix scaffolds. Tissue Eng Part A. 2009 May;15(5):1119-25. doi: 10.1089/ten.tea.2008.0162. PMID 18837648
- [Background] Holcomb JB, Stansbury LG, Champion HR, Wade C, Bellamy RF. Understanding combat casualty care statistics. J Trauma. 2006 Feb;60(2):397-401. doi: 10.1097/01.ta.0000203581.75241.f1. PMID 16508502
- [Background] Mazurek MT, Ficke JR. The scope of wounds encountered in casualties from the global war on terrorism: from the battlefield to the tertiary treatment facility. J Am Acad Orthop Surg. 2006;14(10 Spec No.):S18-23. doi: 10.5435/00124635-200600001-00005. PMID 17003195
- [Background] Noe A. Extremity injury in war: a brief history. J Am Acad Orthop Surg. 2006;14(10 Spec No.):S1-6. doi: 10.5435/00124635-200600001-00002. PMID 17003177
- [Background] Hostetler SG, Schwartz L, Shields BJ, Xiang H, Smith GA. Characteristics of pediatric traumatic amputations treated in hospital emergency departments: United States, 1990-2002. Pediatrics. 2005 Nov;116(5):e667-74. doi: 10.1542/peds.2004-2143. PMID 16263981
- [Background] Crisan M, Yap S, Casteilla L, Chen CW, Corselli M, Park TS, Andriolo G, Sun B, Zheng B, Zhang L, Norotte C, Teng PN, Traas J, Schugar R, Deasy BM, Badylak S, Buhring HJ, Giacobino JP, Lazzari L, Huard J, Peault B. A perivascular origin for mesenchymal stem cells in multiple human organs. Cell Stem Cell. 2008 Sep 11;3(3):301-13. doi: 10.1016/j.stem.2008.07.003. PMID 18786417
- [Background] Reing JE, Zhang L, Myers-Irvin J, Cordero KE, Freytes DO, Heber-Katz E, Bedelbaeva K, McIntosh D, Dewilde A, Braunhut SJ, Badylak SF. Degradation products of extracellular matrix affect cell migration and proliferation. Tissue Eng Part A. 2009 Mar;15(3):605-14. doi: 10.1089/ten.tea.2007.0425. PMID 18652541
- [Background] Zantop T, Gilbert TW, Yoder MC, Badylak SF. Extracellular matrix scaffolds are repopulated by bone marrow-derived cells in a mouse model of achilles tendon reconstruction. J Orthop Res. 2006 Jun;24(6):1299-309. doi: 10.1002/jor.20071. PMID 16649228
- See also: Musclotendinous Tissue Repair Unit and Reinforcement (MTURR) — http://clinicaltrials.gov